CLINICAL TRIAL: NCT00367549
Title: Nutrition as Determinant of Labor Outcome
Brief Title: Nutrition as a Determinant of Labor Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Kristin Kardel, Stip., Rikshospitalet University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REK-SØR: S-05308
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2010-05

CONDITIONS: Labor, Obstetric
Keywords: Labor; instrumental delivery; nutrition; epidural anesthesia; oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Dietary Supplement: Energy-containing soft drink — Commercial energy/sports drink

SUMMARY:
This is a randomized, double-blind trial looking at how nutrition intake is associated with labor progress and complications.

DETAILED DESCRIPTION:
Insufficient intake of energy during labor may result in poor labor progress. The study investigates the effect of an energy supplement during labor.

ELIGIBILITY:
Inclusion Criteria:

* Women at gestational age > 36 weeks, parity 0

Exclusion Criteria:

* Gestational age < 36 weeks
* Signs of fetal pathology:

  * Different or abnormal (pathological) CTG test performed just before start of the test
  * Abnormal Doppler registrations (PI in the arteria umbilicae > 2SD for the gestational age)
  * Established notch in the arteria uterinae or notch bilaterally or PI > 2SD > 24 weeks
  * Diverging in the weight of the fetus > - 22% or diverging in the growth of the fetus - 10% or more, and established structural pathology in the fetus, oligohydramnion (amniotic fluid index < 6)
* Maternal diseases and pregnancy complications

  * diabetes in pregnancy
  * high blood pressure
  * cardiovascular diseases
  * rheumatic disease
  * epilepsia
  * lung disease, etc.

CTG test: cardiotocographic test (a measure of fetal activity)

PI: pulsatory index (velocity pattern)

SD: standard deviation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The course of the labor by women (parity 0) at gestational age > 36 weeks, including: total labor time | At time of birth

SECONDARY OUTCOMES:
Length of stage 1 (cervical opening < 10 cm) and stage 2 (pushing time)
Use of epidural anesthetics
Use of contraction-stimulating drugs
Instrumental delivery

CONTACTS AND LOCATIONS:
Overall Officials: Tore Henriksen, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Kristin Kardel, Oslo, Norway